CLINICAL TRIAL: NCT03077204
Title: Clinical and Radiographic Outcomes of BIO4 Bone Matrix in Patients Undergoing 1 or 2-Level Anterior Cervical Discectomy and Fusion Surgery
Brief Title: BIO4 Clinical Case Study: Cervical Spine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seton Healthcare Family (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-16-109
Record Dates: First submitted 2017-02-27; First posted 2017-03-10 (Actual); Results first posted 2022-01-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Degenerative Disc Disease; Trauma (Including Fractures); Spondylolisthesis
Keywords: Total cervical vertebrectomy; Partial cervical vertebrectomy; Failed previous fusion; Spinal stenosis; Tumor; Decompression of the spinal cord; Pseudoarthrosis; Curvatures; Deformities
MeSH Terms: conditions — Intervertebral Disc Degeneration; Wounds and Injuries; Spondylolisthesis; Spinal Stenosis; Neoplasms; Pseudarthrosis; Congenital Abnormalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- BIO4 treatment (Other): Patients undergoing 1 or 2-level Anterior Cervical Discectomy and Fusion (ACDF) spine surgery utilizing BIO4 with Bio AVS Cervical Allograft (with graft window).
  Interventions: Biological: 1 or 2-Level ACDF utilizing BIO4 with Bio AVS Cervical Allograft (with graft window).; Device: Aviator Anterior Cervical Plating System

INTERVENTIONS:
Biological: 1 or 2-Level ACDF utilizing BIO4 with Bio AVS Cervical Allograft (with graft window). — The study will utilize the BIO4 on label as a 361 HCT/P (human cell, tissue and cellular and tissue-based product) for homologous use for the repair, replacement or reconstruction of bone defects. Interbody fusion (1 or 2-level fusion) in conjunction with an allograft (hct/p) interbody spacer (anterior approach in the cervical spine with hardware). Investigators will also use the Aviator Anterior Cervical Plating System for anterior intervertebral screw fixation of the cervical spine at levels C2-T1. The Aviator Anterior Cervical Plating System is intended for use as an aid in cervical spinal fusion and is intended for unilateral fixation. The Aviator plates are intended to be used with the Aviator bone screws.
Device: Aviator Anterior Cervical Plating System — The study will utilize the BIO4 on label as a 361 HCT/P (human cell, tissue and cellular and tissue-based product) for homologous use for the repair, replacement or reconstruction of bone defects. Interbody fusion (1 or 2-level fusion) in conjunction with an allograft (hct/p) interbody spacer (anterior approach in the cervical spine with hardware). Investigators will also use the Aviator Anterior Cervical Plating System for anterior intervertebral screw fixation of the cervical spine at levels C2-T1. The Aviator Anterior Cervical Plating System is intended for use as an aid in cervical spinal fusion and is intended for unilateral fixation. The Aviator plates are intended to be used with the Aviator bone screws.

SUMMARY:
The goal of this study is to investigate the efficacy of BIO4 bone matrix in patients undergoing 1 or 2-level Anterior Cervical Discectomy and Fusion (ACDF) spine surgery. Specifically, the study aims to collect the data for ACDF model utilizing BIO4 with Bio AVS Cervical Allograft (with graft window).

DETAILED DESCRIPTION:
This is a prospective study with the intent to investigate the efficacy of BIO4 bone matrix in patients undergoing 1 or 2-level Anterior Cervical Discectomy and Fusion (ACDF) spine surgery. At the time a patient is scheduled for surgery, the patient's chart will be evaluated for inclusion/exclusion criteria. If a patient meets the criteria for the study, the study will be explained to the patient and consent obtained.

Investigators will utilize the BIO4 on label as a 361 HCT/P (human cell, tissue and cellular and tissue-based product) for homologous use for the repair, replacement or reconstruction of bone defects. Interbody fusion (1 or 2-level fusion) in conjunction with an allograft (hct/p) interbody spacer (anterior approach in the cervical spine with hardware) will be utilized.

Investigators will also use the Aviator Anterior Cervical Plating System for anterior intervertebral screw fixation of the cervical spine at levels C2-T1. The Aviator Anterior Cervical Plating System is intended for use as an aid in cervical spinal fusion and is intended for unilateral fixation. The Aviator plates are intended to be used with the Aviator bone screws.

Study Outcomes:

* Radiological assessment (cervical spine x-ray and if needed, computed tomography (CT) at 1 year follow up)of fusion as the primary endpoint
* Arthrodesis rates assessed using CT (1 year follow up, if needed) and Anterior-Posterior (AP), lateral and dynamic flexion-extension cervical spine x-rays pre-operative (pre-op), post-operatively (post-op) 2~4 weeks (10~34 days post op), 3 months (83~97 days post-op), 6 months (173~187 days post-op) and 1 year post-op (351~379 days post op, primary data point outcome)
* Revision rates
* Outcome scores: Visual Analog Scale (VAS) and Neck Disability Index (NDI) pre-op, post-op 2~ 4weeks, 3 months, 6 months and 1 year.

The null hypothesis is that in ACDF model, the clinical and radiographic outcomes of utilizing BIO4 bone matrix with Bio AVS Cervical Allograft are equivalent to historical high level published data of similar product (Data reported in Meta-analysis ACDF obtained from FDA disc arthroplasty trials).

ELIGIBILITY:
Inclusion Criteria

1. Age>18 years
2. Scheduled 1 or 2-level ACDF spine surgery
3. The capacity to provide informed consent.
4. Subject has one or more of the following diagnoses:

   1. Degenerative Disc Disease (as defined by neck pain of discogenic origin with degeneration of the disc confirmed by patient history and radiographic studies)
   2. Trauma (including fractures)
   3. Tumors
   4. Deformities or curvatures (including kyphosis, lordosis, or scoliosis)
   5. Pseudoarthrosis
   6. Failed previous fusion
   7. Decompression of the spinal cord following total or partial cervical vertebrectomy
   8. Spondylolisthesis
   9. Spinal stenosis

Exclusion Criteria Patients with any of the following conditions will be excluded, or if enrolled and found to be ineligible and do not fit the inclusion criteria, will be withdrawn from the study.

1. Patients with current or recent history of malignancy or infectious disease.
2. The inability to provide informed consent.
3. Subject has marked local inflammation
4. Subject has any mental or neuromuscular disorder which would create an unacceptable risk of fixation failure or complications in postoperative care.
5. Subject has a bone stock compromised by disease, infection or prior implantation which cannot provide adequate support and/or fixation to the devices.
6. Subject has bone abnormalities preventing safe screw fixation.
7. Subject has any open wounds.
8. Subject has rapid joint disease, bone absorption, osteopenia, osteomalacia, and/or osteoporosis. Osteoporosis or osteopenia are relative contraindications, since this condition may limit the degree of obtainable correction and/or the amount of mechanical fixation.
9. Subject has a documented or suspected metal sensitivity.
10. Subject is pregnant.
11. Subject has anatomical structures or physiological performance that would interfere with implant utilization.
12. Subject has inadequate tissue coverage over the operative site.
13. Subject has other medical or surgical conditions which would preclude the potential benefit of surgery, such as congenital abnormalities, immunosuppressive disease, elevation of sedimentation rate unexplained by other diseases, elevation of white blood count (WBC), or marked left shift in the WBC differential count.
14. Note: The Aviator Anterior Cervical Plating System is not approved or intended for screw attachment to the posterior elements (pedicles) of the cervical, thoracic, or lumbar spine. The surgeon must consider the levels of implantation, patient weight, patient activity level, and other patient conditions which may impact on the performance of the system.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eeric Truumees, MD, Principal Investigator — Seton Spine and Scoliosis Center
Locations (1):
- Seton Spine and Scoliosis Center, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roberts TT, Rosenbaum AJ. Bone grafts, bone substitutes and orthobiologics: the bridge between basic science and clinical advancements in fracture healing. Organogenesis. 2012 Oct-Dec;8(4):114-24. doi: 10.4161/org.23306. Epub 2012 Oct 1. PMID 23247591
- [Background] • Osiris Therapeutics-Data on File
- [Background] • Bourke HE, Sandison A, Hughes SPF and Reichert ILH. Vascular Endothelial Growth Factor (VEGF) in Human Periosteum- Normal Expression and Response to Fracture, "Journal of Bone and Joint Surgery, British Volume (2003)
- [Background] Epstein NE. An analysis of noninstrumented posterolateral lumbar fusions performed in predominantly geriatric patients using lamina autograft and beta tricalcium phosphate. Spine J. 2008 Nov-Dec;8(6):882-7. doi: 10.1016/j.spinee.2007.11.005. Epub 2008 Feb 14. PMID 18280215
- [Background] Epstein NE. Beta tricalcium phosphate: observation of use in 100 posterolateral lumbar instrumented fusions. Spine J. 2009 Aug;9(8):630-8. doi: 10.1016/j.spinee.2009.04.007. Epub 2009 Jun 4. PMID 19501025
- [Background] Eastlack RK, Garfin SR, Brown CR, Meyer SC. Osteocel Plus cellular allograft in anterior cervical discectomy and fusion: evaluation of clinical and radiographic outcomes from a prospective multicenter study. Spine (Phila Pa 1976). 2014 Oct 15;39(22):E1331-7. doi: 10.1097/BRS.0000000000000557. PMID 25188591

RESULTS

PARTICIPANT FLOW:
Groups:
- BIO4 Treatment: Participants were treated as per the protocol.
Period: Overall Study
Arm/Group | BIO4 Treatment
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- BIO4 Treatment: Treatment group consisted of patient undergoing ACDF using BIO4
Arm/Group | BIO4 Treatment
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 4
Age, Continuous [Mean (Full Range); unit: years] | 57.4 [45 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Visual Analog Scale [Mean (Full Range); unit: units on a scale] — Range: 0-10 0= no pain 10= worst pain
  units on a scale | 4.7 [0 to 8]
Neck Disability Index [Mean (Full Range); unit: units on a scale] — 0-100 (0=better, 100=worst)
  units on a scale | 35 [6 to 68]

OUTCOME MEASURES:

1. Primary Outcome: Radiological Assessment : Fusion Status
Description: This will be used to monitor the fusion status at 1 year post-op. The fusion states was reported as the number of patients who fused. If fused, then we say "Yes". We counted the number of patients who fused. If all 20 patients fused then we said there were 20 "yes".
Time Frame: Post-op 1 year
Population: Patients who underwent ACDF using BIO4
Measure: Number; unit: participants
Groups:
- BIO4 Treatment: Patients undergoing ACDF using BIO4
Arm/Group | BIO4 Treatment
Number analyzed (Participants) | 20
participants | 20

2. Primary Outcome: Arthrodesis Rates
Description: Anterior-Posterior (AP), lateral and dynamic flexion-extension cervical spine x-rays will be used to access arthrodesis rates at different time intervals. We counted the number of patients who developed arthrodesis. The arthrodesis rate was calculated as the number of patients who developed arthrodesis.
Time Frame: Post-op 1 year
Population: Patients who underwent ACDF using BIO4
Measure: Number; unit: participants
Arm/Group | BIO4 Treatment
Number analyzed (Participants) | 20
participants | 0

3. Secondary Outcome: Revision Rates (if Any)
Description: As needed, any post-operative surgical revision rates will be accessed. The revision rate was described as the number of patients who had to undergo revision post index surgery
Time Frame: Post-op 2~4 weeks
Population: Patients who underwent ACDF using BIO4
Measure: Number; unit: participants
Arm/Group | BIO4 Treatment
Number analyzed (Participants) | 20
participants | 0

4. Secondary Outcome: Revision Rates (if Any)
Description: as for outcome 3
Time Frame: Post-op 3 months
Population: Patients who underwent ACDF using BIO4
Measure: Number; unit: participants
Arm/Group | BIO4 Treatment
Number analyzed (Participants) | 20
participants | 0

5. Secondary Outcome: Revision Rates (if Any)
Description: as for outcome 3
Time Frame: Post-op 6 months
Population: Patients who underwent ACDF using BIO4
Measure: Number; unit: participants
Arm/Group | BIO4 Treatment
Number analyzed (Participants) | 20
participants | 0

6. Secondary Outcome: Revision Rates (if Any)
Description: as for outcome 3
Time Frame: Post-op 1 year
Population: Patients who underwent ACDF using BIO4
Measure: Number; unit: participants
Arm/Group | BIO4 Treatment
Number analyzed (Participants) | 20
participants | 0

7. Secondary Outcome: VAS
Description: Patient reported VAS will be collected at different time intervals. The revision rate was described as the number of patients who had to undergo revision post index surgery. VAS: 0-10 (0=better, 10=worst)
Time Frame: Pre-op
Population: Patients treated with BIO4
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | BIO4 Treatment
Number analyzed (Participants) | 20
units on a scale | 4.7 [0 to 8]

8. Secondary Outcome: VAS
Description: Patient reported VAS will be collected at different time intervals. VAS: 0-10 (0=better, 10=worst)
Time Frame: Post-op 2 ~ 4 weeks
Population: Patients who underwent ACDF using BIO4
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | BIO4 Treatment
Number analyzed (Participants) | 20
units on a scale | 2.9 [0 to 7]

9. Secondary Outcome: VAS
Description: Patient reported VAS will be collected at different time intervals. VAS: 0-10 (0=better, 10=worst)
Time Frame: Post-op 3 months
Population: Patients who underwent ACDF using BIO4
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | BIO4 Treatment
Number analyzed (Participants) | 20
units on a scale | 2.4 [0 to 7]

10. Secondary Outcome: VAS
Description: Patient reported VAS will be collected at different time intervals. VAS: 0-10 (0=better, 10=worst)
Time Frame: Post-op 6 months
Population: Patients who underwent ACDF using BIO4
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | BIO4 Treatment
Number analyzed (Participants) | 20
units on a scale | 2 [0 to 5]

11. Secondary Outcome: VAS
Description: Patient reported VAS will be collected at different time intervals. VAS: 0-10 (0=better, 10=worst)
Time Frame: Post-op 1 year
Population: Patients who underwent ACDF using BIO4
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | BIO4 Treatment
Number analyzed (Participants) | 20
units on a scale | 1.2 [0 to 6]

12. Secondary Outcome: NDI
Description: Patient reported NDI will be collected at different time intervals. NDI: 0-100 (0=better, 100=worst)
Time Frame: Pre-op
Population: Patients who underwent ACDF using BIO4
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | BIO4 Treatment
Number analyzed (Participants) | 20
units on a scale | 35 [6 to 68]

13. Secondary Outcome: NDI
Description: Patient reported NDI will be collected at different time intervals NDI: 0-100 (0=better, 100=worst)
Time Frame: Post-op 2~4 weeks
Population: Patients who underwent ACDF using BIO4
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | BIO4 Treatment
Number analyzed (Participants) | 20
units on a scale | 19.1 [8 to 60]

14. Secondary Outcome: NDI
Description: Patient reported NDI will be collected at different time intervals. NDI: 0-100 (0=better, 100=worst)
Time Frame: Post-op 3 months
Population: Patients who underwent ACDF using BIO4
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | BIO4 Treatment
Number analyzed (Participants) | 20
units on a scale | 20.7 [0 to 48]

15. Secondary Outcome: NDI
Description: Patient reported NDI will be collected at different time intervals. NDI: 0-100 (0=better, 100=worst)
Time Frame: Post-op 6 months
Population: Patients who underwent ACDF using BIO4
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | BIO4 Treatment
Number analyzed (Participants) | 20
units on a scale | 18.7 [0 to 58]

16. Secondary Outcome: NDI
Description: Patient reported NDI will be collected at different time intervals. NSI: 0-100 (0=better, 100=worst)
Time Frame: Post-op 1 year
Population: Patients who underwent ACDF using BIO4
Measure: Mean (Full Range); unit: units on a scale
Groups:
- BIO4 Treatment: 9.1±2.4(0-36)
Arm/Group | BIO4 Treatment
Number analyzed (Participants) | 20
units on a scale | 9.1 [0 to 36]

17. Secondary Outcome: Arthrodesis Rates
Description: Anterior-Posterior (AP), lateral and dynamic flexion-extension cervical spine x-rays will be used to access arthrodesis rates at different time intervals. The arthrodesis rate was calculated as the number of patients who developed arthrodesis.
Time Frame: Pre-op
Population: Patients who underwent ACDF using BIO4
Measure: Number; unit: participants
Arm/Group | BIO4 Treatment
Number analyzed (Participants) | 20
participants | 0

18. Secondary Outcome: Arthrodesis Rates
Description: as for outcome 17
Time Frame: Post-op 2~4 weeks
Population: Patients who underwent ACDF using BIO4
Measure: Number; unit: participants
Arm/Group | BIO4 Treatment
Number analyzed (Participants) | 20
participants | 0

19. Secondary Outcome: Arthrodesis Rates
Description: as for outcome 17
Time Frame: Post-op 3 months
Population: Patients who underwent ACDF using BIO4
Measure: Number; unit: participants
Arm/Group | BIO4 Treatment
Number analyzed (Participants) | 20
participants | 0

20. Secondary Outcome: Arthrodesis Rates
Description: as for outcome 17
Time Frame: Post-op 6 months
Population: Patients who underwent ACDF using BIO4
Measure: Number; unit: participants
Arm/Group | BIO4 Treatment
Number analyzed (Participants) | 20
participants | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: We reviewed mortality in all our 20 patients
Arm/Group | BIO4 Treatment
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 1/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIO4 Treatment (N=20)
Sepsis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIO4 Treatment (N=20)
Respiratory distress post-surgery (Surgical and medical procedures) | 1 (1) — Patient re-intubated for respiratory distress post-surgery

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-28): https://cdn.clinicaltrials.gov/large-docs/04/NCT03077204/Prot_SAP_001.pdf